CLINICAL TRIAL: NCT04305158
Title: Colonoscopy Using Nitrous Oxide- A Pilot Study in the USA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 239435
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Nitrous Oxide
Keywords: Moderate sedation; Nitrous oxide; Screen colonoscopy
MeSH Terms: interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrous Oxide (Experimental): Patient receiving Nitrous Oxide are evaluated for success of the procedure
  Interventions: Drug: Nitrous Oxide
- IV Sedation group (Active Comparator): In this group a combination of Midazolam and Fentanyl is used per endoscopic discretion
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous Oxide — Patient receiving nitrous oxide are evaluated for success of the procedure

SUMMARY:
Colon cancer is the second most common cancer in men and the third most common cancer in women worldwide. The clinical objectives of administering sedation for GI endoscopy are to relieve patient anxiety and discomfort and to improve the outcome of the examination. Use of N2O could potentially provide an alternate safe and cheap option for patients who do not prefer IV sedation for colonoscopy

DETAILED DESCRIPTION:
Patients who are considered low risk for anesthesia administration (ASA class <IV) receive moderate sedation with a combination of intravenous benzodiazepine and opioid medication. an alternative method of providing analgesia with "on-demand" inhalation of nitrous oxide (hereafter referred to as N2O) combined with oxygen has been postulated. Nitrous Oxide has been used for analgesia in various procedures including childbirth, general anesthesia, pediatric dentistry, bone marrow aspiration, fracture reductions, and minor surgical procedures (surgical dressings, pulmonary endoscopy, an abscess . It could potentially reduce overall costs for the procedure, in addition to providing a quicker recovery, turn over

ELIGIBILITY:
Inclusion Criteria:

Men and women, more than 18 years old Scheduled for a colonoscopy at the Endoscopy unit

Exclusion Criteria:

* High ASA risk (IV/ >)
* History of chronic pain
* Allergy to N2O or opioid or BDZ
* No consent
* Recent head injury with impairment of consciousness or Intracranial / Middle Ear surgery within the previous 6 months with or without residual deficits.
* Pneumothorax, air embolism
* Decompression sickness or within 48 hours of an underwater dive
* Severe emphysema with bullae
* Gross abdominal distension with suspicion for bowel obstruction
* Intoxication
* Maxillofacial injuries (where patient unable to administer the drug using a mouthpiece/mask, or there is the risk of causing further damage to facial wounds and there may also be a significant risk of blood inhalation)
* Patients with chronic pulmonary disease for whom an inspired oxygen concentration of more than 28% oxygen might be dangerous
* Patients on Methotrexate
* Where patients need assistance to hold the mask or mouthpiece.
* Retinal surgery within the last three months
* Any patient who does not otherwise clinically qualify for standard sedation methods (i.e., those who require general anesthesia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Cecal intubation rates and time of the procedure - total time and recovery | 1 to 30 minutes
  Time required to complete the procedure and reach end of the colon

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Dehmel, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States